CLINICAL TRIAL: NCT00632021
Title: Pharmacist Intervention for Low-Literacy in Cardiovascular Disease
Brief Title: Pharmacist Intervention to Decrease Medication Errors in Heart Disease Patients (The PILL-CVD Study)
Acronym: PILL-CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sunil Kripalani, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 539; R01HL089755 (NIH)
Record Dates: First submitted 2008-03-06; First posted 2008-03-10 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome; Heart Failure
Keywords: Low Health Literacy; Medication Errors; Cardiovascular Disease; Pharmacist; Care Transition
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Patients will receive usual care at hospital discharge, which generally includes physician reconciliation of medications and a nurse-provided explanation of how to take medications at the time of discharge.
- 2 (Experimental): Participants will receive pharmacist-led medication reconciliation, pharmacist counseling prior to discharge, a follow-up telephone call 1-4 days after discharge, and additional telephone support as needed.
  Interventions: Behavioral: Pharmacist Intervention for Low-Literacy in Cardiovascular Disease

INTERVENTIONS:
Behavioral: Pharmacist Intervention for Low-Literacy in Cardiovascular Disease — Before hospital discharge, a pharmacist will provide medication reconciliation and counseling on how to take medications. Participants will receive a follow-up phone call 1 to 4 days after hospital discharge to discuss any medication problems, and additionally as needed.
  Arms: 2

SUMMARY:
Many people who have recently left the hospital have difficulties managing their medications, and medication errors are common. Patients with low health literacy levels may have a particularly difficult time understanding medication dosing and instructions. This study will evaluate a literacy-focused program that provides educational assistance from pharmacists at the time of hospital discharge to people hospitalized with heart problems.

DETAILED DESCRIPTION:
After hospital discharge, many people experience difficulty in managing their medication regimens. This can be due to medication dosing changes, challenges in adjusting new medications with those that were taken previously, inadequate discharge instructions from hospital personnel, and inadequate follow-up. Difficulty with medication management can lead to medication errors that result in harmful side effects, poor disease control, hospital readmission, or even death. People with low health literacy often have greater difficulty with understanding and managing their medication regimens and as a result they experience more medication use errors. Although research shows that many medication errors could be prevented or lessened through improved doctor communication and patient-centered treatment programs, little research has been done on the effectiveness of such programs among low-literacy patients or of such programs during key transition times like hospital discharge. Getting pharmacists involved with patient care before hospital discharge may prevent unnecessary and dangerous medication errors from occurring once patients leave the hospital. Because of the severity of heart conditions and the likelihood of serious adverse effects from non-compliance with heart medications, this study will evaluate people admitted to the hospital for acute coronary syndromes or heart failure. The purpose of this study is to evaluate the effectiveness of a health literacy-focused, pharmacist-delivered program at reducing medication errors in heart patients during the first month after hospital discharge.

This study will enroll people admitted to the hospital who have acute coronary syndromes or heart failure. Participants will be randomly assigned to either the pharmacist-delivered program or usual care. Participants assigned to the intervention group will receive a pharmacist-assisted medication review while in the hospital, counseling from a pharmacist at the time of hospital discharge, a low-literacy education tool that details the discharge medications, a follow-up phone call 1 to 4 days after discharge, and additional phone calls as needed. Participants receiving usual care will receive a doctor-assisted medication review and nurse-provided guidance on medication usage at the time of hospital discharge. Approximately 30 days after hospital discharge, study researchers will call all participants to collect information on serious medication errors, health care utilization, and disease-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating study hospital
* Diagnosis of acute coronary syndromes or heart failure

Exclusion Criteria:

* Too ill to participate
* Corrected visual acuity worse than 20/200
* Severe hearing impairment
* Patient is not being discharged to their home
* No regular telephone number
* Not fluent in English or Spanish
* Unintelligible speech
* In police custody
* Caregiver manages all medications
* Delirium or severe dementia
* Psychotic illness
* Already participating in a conflicting study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kripalani, MD, MSc, Principal Investigator — Vanderbilt University Medical Center; Jeffrey L. Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Schnipper JL, Roumie CL, Cawthon C, Businger A, Dalal AK, Mugalla I, Eden S, Jacobson TA, Rask KJ, Vaccarino V, Gandhi TK, Bates DW, Johnson DC, Labonville S, Gregory D, Kripalani S; PILL-CVD Study Group. Rationale and design of the Pharmacist Intervention for Low Literacy in Cardiovascular Disease (PILL-CVD) study. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):212-9. doi: 10.1161/CIRCOUTCOMES.109.921833. PMID 20233982
- [Result] Kripalani S, Roumie CL, Dalal AK, Cawthon C, Businger A, Eden SK, Shintani A, Sponsler KC, Harris LJ, Theobald C, Huang RL, Scheurer D, Hunt S, Jacobson TA, Rask KJ, Vaccarino V, Gandhi TK, Bates DW, Williams MV, Schnipper JL; PILL-CVD (Pharmacist Intervention for Low Literacy in Cardiovascular Disease) Study Group. Effect of a pharmacist intervention on clinically important medication errors after hospital discharge: a randomized trial. Ann Intern Med. 2012 Jul 3;157(1):1-10. doi: 10.7326/0003-4819-157-1-201207030-00003. PMID 22751755
- [Derived] Bell SP, Schnipper JL, Goggins K, Bian A, Shintani A, Roumie CL, Dalal AK, Jacobson TA, Rask KJ, Vaccarino V, Gandhi TK, Labonville SA, Johnson D, Neal EB, Kripalani S; Pharmacist Intervention for Low Literacy in Cardiovascular Disease (PILL-CVD) Study Group. Effect of Pharmacist Counseling Intervention on Health Care Utilization Following Hospital Discharge: A Randomized Control Trial. J Gen Intern Med. 2016 May;31(5):470-7. doi: 10.1007/s11606-016-3596-3. PMID 26883526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults admitted to Vanderbilt University Hospital or Brigham and Women's Hospital for acute coronary syndromes or acute decompensated heart failure were enrolled between May 2008 and September 2009. We enrolled and randomized 862 patients. Eleven patients withdrew consent or died in the hospital, leaving 851 patients in the analysis.
Pre-assignment Details: This was a randomized, controlled trial with concealed allocation and blinded outcome assessors. We enrolled and randomized 862 patients (430 intervention and 432 usual care). Eleven patients (7 intervention and 4 usual care) withdrew consent or died in the hospital, leaving 851 patients in the intention-to-treat analysis.
Groups:
- Control (Usual Care): Control (usual care) arm
- Intervention: Intervention arm
Period: Overall Study
Arm/Group | Control (Usual Care) | Intervention
Started | 432 | 430
Completed | 428 | 423
Not Completed | 4 | 7
Not completed — Withdrawal/death | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Usual Care) | Intervention | Total
Number analyzed (Participants) | 428 | 423 | 851
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14) | 61 (14) | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 173 | 352
  Male | 249 | 250 | 499
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 71 | 77 | 148
  White | 335 | 319 | 654
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 21 | 37
Region of Enrollment [Number; unit: Number of participants]
  United States | 428 | 423 | 851
Study Site [Count of Participants; unit: Participants]
  Vanderbilt University Hospital | 200 | 197 | 397
  Brigham and Women's Hospital | 228 | 226 | 454
Health literacy (sTOFHLA score) [Count of Participants; unit: Participants] — Short Test of Functional Health Literacy in Adults
  Participants
    Inadequate | 39 | 47 | 86
    Marginal | 38 | 36 | 74
    Adequate | 340 | 331 | 671
    Missing | 11 | 9 | 20
Language [Count of Participants; unit: Participants]
  English | 425 | 414 | 839
  Spanish | 3 | 9 | 12
Education [Median (Inter-Quartile Range); unit: years] | 14 [12 to 16] | 14 [12 to 16] | 14 [12 to 16]
Income [Count of Participants; unit: Participants]
  <10K | 17 | 20 | 37
  10K to <15K | 24 | 21 | 45
  15K to <20K | 19 | 23 | 42
  20K to <25K | 47 | 56 | 103
  25K to <35K | 49 | 49 | 98
  35K to <50K | 56 | 54 | 110
  50K to <75K | 60 | 58 | 118
  75K+ | 119 | 105 | 224
  Missing | 37 | 37 | 74
Cognition (Mini cog score) [Count of Participants; unit: Participants]
  Impaired | 46 | 52 | 98
  Not impaired | 380 | 371 | 751
  Missing | 2 | 0 | 2
Has primary care provider [Count of Participants; unit: Participants]
  Yes | 392 | 386 | 778
  No | 36 | 37 | 73
Number of pre-admission medications [Median (Inter-Quartile Range); unit: Medications] | 7 [4 to 11] | 8 [4 to 11] | 8 [4 to 11]
Comorbidities [Number; unit: participants]
  Diabetes | 195 | 140 | 335
  Hypertension | 296 | 306 | 602
  Hypercholesterolemia | 236 | 234 | 470
  Coronary artery disease | 211 | 225 | 436
  Prior myocardial infarction | 73 | 100 | 173
  Prior stroke or cerebrovascular event | 41 | 30 | 71
  Prior coronary revascularization procedure | 195 | 203 | 398
Marital status [Count of Participants; unit: Participants]
  Married/cohabitating | 256 | 226 | 482
  Single/living alone | 172 | 197 | 369
Insurance status [Count of Participants; unit: Participants]
  Medicare | 162 | 177 | 339
  Medicaid | 37 | 44 | 81
  Commercial | 203 | 167 | 370
  Self-pay/other | 26 | 35 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Medication Errors as Determined by Interview and Medical Chart Review
Description: Number of clinically important medication errors per patient
Time Frame: Measured at Day 30
Measure: Mean (Standard Deviation); unit: serious medication errors
Groups:
- Control: Control (usual care) arm
Arm/Group | Control | Intervention
Number analyzed (Participants) | 428 | 423
serious medication errors | 0.95 (1.36) | 0.87 (1.18)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Equivalence — In the primary analysis we compared the number of clinically important medication errors by treatment group using unadjusted negative binomial regression; Incidence Rate Ratio (IRR) = 0.92, 95% CI 2-sided [0.77 to 1.09]

2. Secondary Outcome: Number of Participants With Unplanned Hospitalizations and Emergency Department Visits
Description: Unplanned hospitalizations and Emergency Department visits
Time Frame: Measured at Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Usual Care) | Intervention
Number analyzed (Participants) | 428 | 423
Participants
  Hospital readmission | 66 | 61
  No readmission | 362 | 362
Statistical Analysis 1: Comparison: Control (Usual Care) vs Intervention; Test type: Equivalence — The association between intervention and time to first unplanned health care event (hospital readmission) was examined using multivariable Cox proportional hazards regression models; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.63 to 1.28]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Any adverse events related to study participation were collected by researchers and reported to the IRB appropriately.
Arm/Group | Control (Usual Care) | Intervention
All-Cause Mortality (participants affected / at risk) | 0/428 | 0/423
Serious Adverse Events (participants affected / at risk) | 0/428 | 0/423
Other Adverse Events (participants affected / at risk) | 0/428 | 0/423

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No